CLINICAL TRIAL: NCT07074275
Title: Predictive Relationship Between Chronic Fibromyalgia Pain and Lifestyle Factors and Role of Inflammation: A Pilot Trial
Brief Title: Chronic Fibromyalgia Pain, Lifestyle Factors, and Inflammation
Acronym: BUFS
Status: Active, not recruiting | Type: Observational
Sponsor: Bournemouth University (Other)
Collaborators: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Omer Elma, Lecturer, Bournemouth University
Other Study IDs: 61104
Record Dates: First submitted 2025-06-30; First posted 2025-07-20 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Fibromyalgia (FM)
Keywords: Fibromyalgia; Chronic musculoskeletal pain; lifestyle; inflammation; Fitbit; Quantitative sensory testing; Physical activity; sleep; Diet; temporal summation; conditioned pain modulation; IL-6; IL-10; TNF-alpha
MeSH Terms: conditions — Fibromyalgia; Inflammation; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum inflammatory biomarkers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to understand how lifestyle factors (such as diet, physical activity, sleep, stress, smoking, and alcohol intake) predict changes in pain sensitivity and modulation in adults aged 18-65 with chronic fibromyalgia pain. The main questions it aims to answer are:

What is the predictive relationship between lifestyle factors and pain sensitivity/modulation? What is the mediating role of inflammation in the relationship between lifestyle factors and pain?

Researchers will explore how various lifestyle factors collectively and individually relate to pain responses and whether inflammatory markers (IL-6, TNF-α, IL-10) mediate these associations.

Participants will:

Wear a Fitbit for two weeks to measure physical activity and sleep Use the Nutritics app to log food intake Complete an online questionnaire on pain, sleep quality, stress, and quality of life Undergo pain sensitivity testing using a digital algometer and pressure cuff Have body weight, height, and BMI measured Provide a blood sample for analysis of inflammatory markers via ELISA

DETAILED DESCRIPTION:
Chronic fibromyalgia pain is a complex and multifaceted condition that significantly affects quality of life and daily functioning. Despite its high prevalence and burden, effective long-term treatment options remain limited. Emerging research highlights the potential influence of modifiable lifestyle factors, such as diet, physical activity, sleep, stress, smoking, and alcohol intake, on pain outcomes, possibly through inflammatory pathways.

This cross-sectional observational study investigates how these lifestyle factors are associated with pain sensitivity and pain modulation mechanisms in adults aged 18 to 65 with a clinical diagnosis of fibromyalgia. It also explores whether systemic inflammation, measured by circulating cytokines (IL-6, TNF-α, and IL-10), mediates these relationships.

Participants will be recruited and screened for eligibility based on age, diagnosis, and health status. Once enrolled, participants will engage in a two-week data collection period during which they will wear a wrist-worn activity tracker (Fitbit) to passively monitor physical activity levels and sleep parameters. Dietary intake will be logged using a mobile nutrition tracking app (Nutritics), and participants will complete validated online questionnaires assessing perceived stress, sleep quality, pain characteristics, and health-related quality of life.

Following the tracking period, participants will attend a clinic session for physiological assessments. Pain sensitivity and modulation will be evaluated using pressure-based methods including a digital algometer and a pressure cuff, both of which are safe and standardized tools in pain research. Anthropometric data, including height, weight, and body mass index (BMI), will be collected using calibrated devices. Finally, a venous blood sample will be drawn for analysis of inflammatory markers using enzyme-linked immunosorbent assay (ELISA).

By examining the interplay between lifestyle factors, inflammatory markers, and pain processing mechanisms, this study aims to generate insights that could inform the development of individualized, non-pharmacological strategies for managing fibromyalgia pain more effectively.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged between 18-65 years old
* Clinically diagnosed with fibromyalgia
* Experiencing chronic musculoskeletal pain for at least 3 months, occurring on a minimum of 3 days per week
* Able to understand study procedures and provide informed consent
* Willing to comply with study requirements (e.g., wear activity tracker, complete food logs, questionnaires, and attend assessment sessions)

Exclusion Criteria:

* Diagnosis of any active cancer or history of cancer within the past 5 years
* Use of immunosuppressive medications (e.g., corticosteroids, chemotherapy, biologics)
* Presence of systemic inflammatory or metabolic conditions, such as: Type 1 or Type 2 Diabetes, Rheumatoid arthritis, Lupus or other autoimmune disorders.
* Current pregnancy or breastfeeding
* Acute infection or illness at the time of data collection
* Inability or unwillingness to comply with study procedures (e.g., technology use, blood draw)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Participants will be selected from the general public, primarily individuals residing in the Dorset area, including Bournemouth, Poole, and Christchurch. Recruitment was conducted through public announcements on social media platforms such as Facebook. The study is open to those who are able and willing to travel to Bournemouth University for in-person assessments. Participants are not limited to any specific clinical setting and represent a community-based sample of adult females diagnosed with fibromyalgia.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2025-08-23 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pressure Pain Threshold | At the second visit (Day 2)
  Pressure pain threshold will be measured with a handheld pressure algometer.
Temporal summation | at the second visit (Day 2)
  Temporal summation will be assessed using a handheld pressure algometer. Following the determination of the individual's pressure pain threshold (PPT), a series of 10 noxious pressure stimuli. The difference in reported pain intensity between the 1st and 10th stimulus application will be calculated as the primary measure of temporal summation.
Conditioned pain modulation | At the second visit (Day 2)
  Conditioned Pain Modulation (CPM) will be assessed using a pressure algometer for the test stimulus and a cuff pressure for the conditioning stimulus. Baseline pressure pain threshold (PPT) will be measured on the dominant trapezius muscle. For the conditioning stimulus, a blood pressure cuff on the non-dominant arm will be inflated and maintained at 200 mmHg, or until the participant reports a pain intensity of 6 out of 10 on a numerical rating scale (NRS), for a duration of 10 minutes. During or immediately following the conditioning stimulus, PPT will be re-measured on the dominant trapezius muscle. The change in PPT from baseline to the conditioning phase will quantify the CPM effect.
Pain Intensity | At the first visit (Day 1)
  Pain intensity will be measured brief pain inventory.
Total sleep duration | between first and second visit.
  Total sleep hours will be measured with Fitbit Charge 6 wearable device.
Sleep Quality | At the first visit (Day 1)
  Sleep quality will be measured with Pittsburg Sleep Quality Index.
Dietary intake | between first and second visit
  Dietary intake will be assessed with 3 day dietary intake dairy. Nutrient intakes will be analysed with use of nutritics software.
Total number of steps | between first and second visit
  Physical activity level will be assessed using data from the Fitbit Charge 6 wearable device, specifically by recording the total number of steps.
Percieved Stress | At the first visit (day 1)
  Perceived stress will be measured using the Perceived Stress Scale (PSS). Scores on the PSS range from 0 to 40, with higher scores indicating greater perceived stress.
Alcohol intake frequency | At the first visit (Day 1)
  Alcohol intake frequency will be assessed by asking participants to select one of seven pre-defined options: 'Daily or almost daily,' 'Three or four times a week,' 'Once or twice a week,' 'One to three times a month,' 'Special occasions only,' 'Never,' or 'Previously'.
Smoking status | At the first visit (Day 1)
  Smoking status will be assessed by asking participants to select one of three pre-defined options: 'Current smoker,' 'Never smoked,' or 'Previous smoker.'

SECONDARY OUTCOMES:
Inflammatory Biomarkers | Baseline assessment
  Serum concentrations of IL-6, TNF-α, and IL-10 as measured by ELISA.
Central sensitization inventory | At the first visit
  Central sensitization will be measured using the Central Sensitization Inventory (CSI). Scores on the CSI range from 0 to 100, with higher scores indicating a greater degree of central sensitization.
Fibromyalgia impact questionnaire | At the first visit (Day 1)
  Fibromyalgia impact will be measured using the Fibromyalgia Impact Questionnaire (FIQ). Scores on the FIQ range from 0 to 100, with higher scores indicating a greater impact of fibromyalgia on daily life.
Body weight | At the second visit (day 2)
  Body weight will be measured using a Seca weight scale and recorded in kilograms (kg).
Body height | At the second visit (Day 2)
  Body height will be measured using a Seca length meter and recorded in centimeters (cm).
Body mass index | at the second visit (day 2)
  weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Locations (1):
- Human Performance Lab, Talbot Campus, Bournemouth University, Bournemouth, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) may be shared with other qualified researchers upon reasonable request, for purposes of secondary analysis or meta-analysis. Data will include raw values for pain sensitivity outcomes, lifestyle measures, and cytokine levels.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: starting from the end of the completion of the study
Access Criteria: Upon reasonable request, by contacting to principal investigator.